CLINICAL TRIAL: NCT07113782
Title: Comparison of Magnesium Sulphate vs Tramadol as Adjuvants in Intrathecal Bupivacaine for Postoperative Pain in TURP Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Armed Forces Institute of Urology, Rawalpindi (Other)
Responsible Party: Principal Investigator, Jawad Ul Hassan, Anaesthesiologist, Armed Forces Institute of Urology, Rawalpindi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Trg 1/RB/2024/008
Record Dates: First submitted 2025-07-16; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Benign Prostatic Hyperplasia Postoperative Pain
Keywords: Magnesium sulphate; Tramadol; Intrathecal anesthesia; Bupivacaine; TURP; Postoperative pain; Hemodynamic stability
MeSH Terms: conditions — Pain, Postoperative | interventions — Magnesium Sulfate; Tramadol

STUDY DESIGN:
Intervention Model Description: This study used a randomized, controlled, parallel assignment interventional model in which participants were allocated into two groups. One group received intrathecal bupivacaine with magnesium sulphate, and the other received bupivacaine with tramadol. The interventions were administered once and compared for postoperative analgesia and hemodynamic stability without crossover.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental - Group M (Magnesium Sulphate) (Experimental): Patients receive 12.5 mg of 0.5% hyperbaric bupivacaine with 50 mg (0.1 mL) magnesium sulphate intrathecally.
  Intervention Name: Magnesium sulphate
  Interventions: Drug: 1. Magnesium Sulphate 2. Tramadol
- Active Comparator - Group T (Tramadol) (Active Comparator): Patients receive 12.5 mg of 0.5% hyperbaric bupivacaine with 25 mg (0.5 mL) tramadol intrathecally.
  Intervention Name: Tramadol
  Interventions: Drug: 1. Magnesium Sulphate 2. Tramadol

INTERVENTIONS:
Drug: 1. Magnesium Sulphate 2. Tramadol — Magnesium Sulphate (Group M): 50 mg magnesium sulphate added to 12.5 mg of 0.5% hyperbaric bupivacaine, administered intrathecally.
  Tramadol (Group T): 25 mg tramadol added to 12.5 mg of 0.5% hyperbaric bupivacaine, administered intrathecally.

SUMMARY:
The goal of this clinical trial is to determine whether adding magnesium sulfate or tramadol to intrathecal bupivacaine improves postoperative pain control and hemodynamic stability in adult male patients undergoing transurethral resection of the prostate (TURP).

The main questions this study aims to answer are:

Does the addition of magnesium sulfate or tramadol prolong the duration of postoperative analgesia compared to bupivacaine alone?

Does either adjuvant provide better intraoperative hemodynamic stability?

Researchers will compare two groups:

One group receiving magnesium sulfate plus bupivacaine

Another group receiving tramadol plus bupivacaine

to see which combination is more effective for pain control and hemodynamic outcomes.

Participants will:

Receive spinal anesthesia with either magnesium sulfate or tramadol added to bupivacaine.

Be monitored during surgery for heart rate, blood pressure, and other vital signs.

Be assessed after surgery for pain levels and time until first request for additional pain medication.

DETAILED DESCRIPTION:
This retrospective, randomized, double-blind clinical trial was conducted to compare the efficacy and safety of magnesium sulfate and tramadol as intrathecal adjuvants to hyperbaric bupivacaine in male patients undergoing transurethral resection of the prostate (TURP) under spinal anesthesia.

The primary aim was to evaluate:

The duration of postoperative analgesia, defined as the time from the completion of surgery to the patient's first request for rescue analgesia.

Intraoperative hemodynamic stability, assessed by monitoring mean arterial pressure, heart rate, and the incidence of hypotension or bradycardia.

A total of 60 adult male patients, aged 50 to 80 years, undergoing elective TURP were randomly allocated into two groups (30 patients each):

Group M (Magnesium Group): Received 12.5 mg of 0.5% hyperbaric bupivacaine with 50 mg of magnesium sulfate intrathecally.

Group T (Tramadol Group): Received 12.5 mg of 0.5% hyperbaric bupivacaine with 20 mg of tramadol intrathecally.

All patients received spinal anesthesia at the L3-L4 or L4-L5 interspace under aseptic conditions. Intraoperative monitoring included ECG, non-invasive blood pressure, and pulse oximetry. Data on hemodynamic parameters were collected at regular intervals throughout the procedure.

Primary Outcome Measures:

Time to first postoperative analgesic request (in minutes)

Mean arterial pressure and heart rate during the procedure

Secondary Outcome Measures:

Time to two-segment regression of the sensory block

Incidence of adverse events including hypotension, bradycardia, nausea, vomiting, pruritus, urinary retention, and respiratory depression

Blinding was maintained for both patients and the investigator recording postoperative outcomes.

The study was conducted in accordance with the ethical standards laid down in the 1964 Declaration of Helsinki and its later amendments. Ethical approval was obtained from the Institutional Review Board of Armed Forces Institute of Urology (AFIU), Rawalpindi. Written informed consent was obtained from all participants prior to inclusion in the study.

This trial was completed before registration and is being submitted retrospectively for transparency and publication compliance.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 50 to 80 years
* Scheduled for elective transurethral resection of the prostate (TURP)
* American Society of Anesthesiologists (ASA) physical status I-II
* Provided written informed consent

Exclusion Criteria:

* Known allergy or hypersensitivity to bupivacaine, tramadol, or magnesium sulfate
* Contraindications to spinal anesthesia (e.g., coagulopathy, infection at the injection site)
* History of chronic opioid use or substance abuse
* Severe hepatic, renal, or cardiac disease
* Neurological or psychiatric disorders affecting pain perception or reporting
* Participation in another clinical trial within the past 30 days

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The study involves TURP (Transurethral Resection of the Prostate), a procedure only performed in male patients.
Enrollment: 60 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Duration of postoperative analgesia | Up to 24 hours postoperatively
  Time (in minutes) from administration of intrathecal drug to the first request for rescue analgesia (VAS ≥ 4).

CONTACTS AND LOCATIONS:
Locations (1):
- AFIU, Rawalpindi, Punjab Province, Pakistan